CLINICAL TRIAL: NCT06677008
Title: Post-market Clinical Follow-up Study Plan for Disposable Endoscopic Linear Cutter Stapler
Status: Not yet recruiting | Type: Observational
Sponsor: Suzhou Kerui Medical Technology Co., Ltd (Other)
Responsible Party: Sponsor
Other Study IDs: CAK-PMCF
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: The Expeditious Transection/resection of Tissues and Creation of Anastomoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Disposable endoscopic linear cutter stapler
  Interventions: Device: Disposable endoscopic linear cutter stapler

INTERVENTIONS:
Device: Disposable endoscopic linear cutter stapler — Investigational devices of all the models of the staplers and its cartridge listed in Study Plan(Plan number: CAK-PMCF)

SUMMARY:
This study conducted a Post-Market Clinical Follow-Up study (PMCF) to evaluate the safety and effectiveness of the disposable endoscopic linear cutter stapler produced by Changzhou Ankang Medical Instrument Co., Ltd., through a retrospective analysis of the clinical data, to evaluate the safety and effectiveness of soft tissue resection, transection and anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Age unlimited and gender unlimited;
* The surgery type shall be endoscopic surgery;
* The departments of surgical procedures: general and thoracic surgical procedures;
* Investigational devices of all the models of the staplers and its cartridge listed in Section 2.3.

Exclusion Criteria:

* Patients undergoing surgery for contraindications to the product, such as severe mucosal edema, non-observation of hemostatic sites for surgery or off-label use, such as liver and spleen;
* Combined with other similar products (stapler) for resection, transection and anastomosis of the surgical site;
* Surgery record is incomplete, unable to extract main indicators related information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For patients who need to be operated for abdominal, gynecologic, pediatric, and thoracic, endoscopic (i.e., endo-therapy) surgery for the expeditious transection/resection of tissues and creation of anastomoses.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Anastomosis success rate | the investigation sites will be collected from January 2023 to September 2024.
  The condition of no reoperation in situ was defined as successful anastomosis as determined by surgical records and hospitalization medical records.

SECONDARY OUTCOMES:
Operation time | The investigation sites will be collected from January 2023 to September 2024.
  Confirmed by surgical records and anesthesia sheets.
Amount of intraoperative blood loss | the investigation sites will be collected from January 2023 to September 2024.
  Confirmed by surgical records/nursing notes.
Intraoperative conversion (caused by the stapler and/or cartridge) | the investigation sites will be collected from January 2023 to September 2024.
  Surgical records confirm the intraoperative conversion, and determine whether the intraoperative conversion is caused by the investigational devices according to the description.
Length of hospitalization | the investigation sites will be collected from January 2023 to September 2024.
  Records were collected for the patient's date of surgery and date of discharge .
  Length of hospitalization(days) = date of discharge - date of surgery
All-cause re-hospitalization rate (within 6 months) | From the date of surgery to six months after the surgery
  Re-hospitalization data of patients within 6 months after surgery were collected.
  Postoperative all-cause re-hospitalization rate = number of all-cause re-hospitalization cases/total cases ×100%

OTHER OUTCOMES:
Adverse events | From the date of surgery to six months after the surgery
  Common adverse events due to the device and treatment were: anastomotic leakage, bleeding, stenosis, fistula, infection, etc.
Device deficiencies | From the date of surgery to six months after the surgery
  Inadequacy of medical device with respect to its identity, quality, durability, reliability, usability, safety or performance.
Serious adverse events | From the date of surgery to six months after the surgery
  Incidence of serious adverse events = Number of serious adverse events/number of enrolled cases ×100%

CONTACTS AND LOCATIONS:
Locations (1):
- Disposable endoscopic linear cutter stapler, Wujin District, Changzhou, China

IPD SHARING:
Plan to Share IPD: No